CLINICAL TRIAL: NCT01468025
Title: A Randomized Double-blind Placebo Study to Determine the Effectiveness of Theramine and a Low Dose Naproxen on the Management of Chronic Back Pain
Brief Title: Effectiveness of Theramine on Chronic Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Targeted Medical Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0708101
Record Dates: First submitted 2011-09-15; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Low Back Pain
Keywords: NSAIDs; Theramine; naproxen; Low back pain; amino acids; CRP; Medical Food
MeSH Terms: conditions — Low Back Pain | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Theramine and naproxen (Active Comparator): Patients in this group were randomly given active Theramine and active naproxen.
  Interventions: Drug: Active Theramine and Active Naproxen
- Theramine and placebo (Active Comparator): Patients in this group were randomly given active Theramine with placebo representing naproxen.
  Interventions: Other: Theramine and naproxen-like placebo
- Naproxen and placebo (Active Comparator): Patients in this group were randomly given active naproxen and placebo to represent Theramine.
  Interventions: Drug: Naproxen and Theramine-like placebo

INTERVENTIONS:
Drug: Active Theramine and Active Naproxen — Co-administration of Theramine and Naproxen, CoPack Kit Theraproxen
  Arms: Theramine and naproxen
Other: Theramine and naproxen-like placebo — Theramine, a medical food, co-administered with naproxen-like placebo
  Arms: Theramine and placebo
Drug: Naproxen and Theramine-like placebo — naproxen co-administered with Theramine-like placebo.
  Arms: Naproxen and placebo

SUMMARY:
This research protocol will compare Theramine to a non-steroidal anti-inflammatory drug (NSAID) in the treatment of chronic back pain. The study will examine the efficacy and tolerability of Theramine alone in patients with chronic back pain in comparison to the NSAID, Naproxen, and the co-administration of Naproxen with Theramine.

DETAILED DESCRIPTION:
After informed consent and screening, volunteers will be entered into a double blind, randomized, three-armed trial, with 40 patients in each group. Patients will receive either Naproxen 250 mg daily, Theramine 2 capsules two times daily, or the co-administration of low-dose Naproxen 250 mg daily with Theramine 2 capsules two times daily for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Back pain lasting greater than six weeks. Pain must be present on at least 5 out of 7 days during each of the two weeks prior to screening visit
2. Analgesic medication used to treat pain at least 4 out of last 7 days and at least 10 days in the last month
3. Men and non-pregnant, non-lactating women over the age of 18 and under the age of 75, able to read, understand and sign English-language informed consent, with diagnosis of back pain and baseline back pain greater than 40 mm out of 100 mm on visual analog scale
4. Those taking an NSAID for pain must discontinue use during a washout period based on the attached five (5) half-lives of drug chart
5. If undergoing physical therapy for back pain, therapy must be stable at least three weeks prior to study and remain the same throughout study
6. If using psychoactive medication which might have analgesic effects, (i.e. anti-depressants or anti-convulsants-), treatment must be stable for at least three months prior to study
7. For men and women of child-bearing potential, must be willing to use adequate contraception and not be pregnant or impregnate their partner during the entire time of study
8. Must be willing to commit to all clinical visits during study-related procedures, including required discontinuation (washout) of analgesic or anti-inflammatory medication prior to Day 1 randomization. The patient must agree to using acetaminophen for rescue medication

Exclusion Criteria:

1. Patients with back surgery in the past six months
2. Patients with significant neurologic impairment, as diagnosed on screening physical examination
3. Patients with evidence or history of fracture of the spine in the past year
4. Patients not fluent in English
5. Use of aspirin for non-arthritic conditions, unless at a dose less than or equal to 325 mg a day, and must be stable for at least one month prior to screening
6. Use of controlled substances and/or opiate analgesic for pain, for more than 5 days within the last 30 days prior to screening visit
7. Receipt of an oral intramuscular or soft-tissue injection of corticosteroid within one month prior to screening
8. Participation in a clinical trial within the one month prior to screening
9. History of epidurals in the past 3 months
10. History of alcohol or substance abuse
11. Uncontrolled or unstable serious cardiovascular, pulmonary, gastrointestinal or urogenital, endocrine, neurologic or psychiatric disorder
12. History of gastrointestinal bleed or documented gastric or duodenal ulcer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Roland-Morris Lower Back Pain Scale | Baseline and Day 28
  The primary efficacy outcome will be the change from baseline in awakening stiffness and pain subscale scores obtained from the Roland-Morris Lower Back Pain Scale.

SECONDARY OUTCOMES:
Oswestry Low Back Pain Scale | Baseline and Day 28
  Change measured in Oswestry low back pain scale.
Visual Analog Scale | Baseline and Day 28
  Change measured in visual analog scale.
Blood Panel | Baseline and Day 28
  Baseline and day 28 blood measurement, CBC, liver panel, CRP.